CLINICAL TRIAL: NCT00256542
Title: A Phase II Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Intravesical Alkalinized Lidocaine-Heparin for the Symptoms of Pelvic Pain and/or Urgency of Bladder Origin
Brief Title: Study of U101 for Bladder Pain and/or Urgency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Urigen (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: URG-101
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Last update posted 2006-09-29 (Estimated); Status verified 2006-08

CONDITIONS: Pelvic Pain; Interstitial Cystitis; Bladder Diseases
Keywords: interstitial cystitis; pelvic pain; urgency; frequency; Pelvic Pain and/or Urgency of Bladder Origin
MeSH Terms: conditions — Pelvic Pain; Cystitis, Interstitial; Urinary Bladder Diseases

INTERVENTIONS:
Drug: Alkalinized Lidocaine-Heparin

SUMMARY:
The purpose of this study is to determine whether intravesical U101 (alkalinized lidocaine-heparin) treatment reduces the symptoms of pelvic pain and/or urgency of bladder origin.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects at least 18 years of age.
* Subjects must have given written informed consent to participate in this trial.
* All female subjects, except those who are post-menopausal and/or surgically sterilized, must consent to use two medically acceptable methods of contraception throughout the entire study period. Medically acceptable methods of contraception that may be used by the subject and/or her partner include: abstinence, birth control pills, diaphragm with spermicide, intrauterine device (IUD), condom and foam, vaginal spermicidal suppository, progestin implant, and Depo-Provera injections.
* Subjects must have had symptoms of pelvic pain and/or urgency.
* Medical history and physical examination results must be clinically acceptable to the Investigator. Medical Monitor may evaluate subjects who don't meet eligibility criteria.
* Female subjects currently using hormone therapy (HT) must have been using HT for at least 3 months.

Exclusion Criteria:

* Subjects less than 18 years of age.
* Subjects with known hypersensitivity to heparin or lidocaine.
* Female subjects who have a positive pregnancy test at the time of screening, who are pregnant or lactating, or who are planning to become pregnant during the study period.
* Subjects who are chronic users of narcotics or who are using any narcotics at the time of study entry.
* Subjects who have hepatic disease or clinically significant abnormal liver function tests (more than twice the upper limit of the normal range).
* Subjects who do not expect to be available for the entire duration of the study.
* Subjects with any coexisting significant medical condition that is likely to interfere with study procedures (cardiovascular, hematological, central nervous system, pulmonary, renal, etc.)
* Subjects who have been treated with dimethyl sulfoxide (DMSO) or other bladder instillation therapies within three months prior to study entry.
* Subjects who have had cystoscopic dilatation of their bladder or urethra within three months of study entry.
* Subjects who have taken or used any investigational drug or device within 30 days before the start of the study, or who are currently enrolled in another investigational study.
* Subjects contemplating having or scheduled for any invasive surgical procedures during the study period.
* Subjects who are unwilling or unable to abide by the requirements of the study.
* History of gastrointestinal (GI) bleeding
* Active bleeding from any source
* Screening activated partial thromboplastin time (aPTT) above normal limits
* Systolic blood pressure (BP) > 180 mmHg or < 90 mmHg at Screening.
* Subjects with an actively bleeding lesion/area in the bladder as detected by urinalysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2006-01; Study Completion 2006-09

PRIMARY OUTCOMES:
Overall improvement in combined symptoms of pain and urgency at 3 weeks

SECONDARY OUTCOMES:
Safety
Reduction in pain on ten point scale at 3 weeks
Reduction in urgency on ten point scale at 3 weeks
Change in number of voids/24 hours
Change in average void volume
Reduction in PUF score (pelvic pain, urgency/frequency) at 3 weeks
Reduction in O'Leary-Sant score at 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: C. Lowell Parsons, MD, Principal Investigator — UCSD
Locations (9):
- United States (9):
  - UCSD Medical Center, San Diego, California
  - Georgia Urology, Cartersville, Georgia
  - St. Mary's Good Samaritan, Centralia, Illinois
  - The Urogynecology Center, Overland Park, Kansas
  - Mid-Michigan Health Centers, Jackson, Michigan
  - Central Park Urology, New York, New York
  - The Urology Center, Greensboro, North Carolina
  - Urologic Specialists of Oklahoma, Inc., Tulsa, Oklahoma
  - Whitmore Urology Office, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Parsons CL. Successful downregulation of bladder sensory nerves with combination of heparin and alkalinized lidocaine in patients with interstitial cystitis. Urology. 2005 Jan;65(1):45-8. doi: 10.1016/j.urology.2004.08.056. PMID 15667861